CLINICAL TRIAL: NCT07141446
Title: Evaluation of Efficacy of Neem (Azadirachta Indica) Versus Triamcinolone Acetonide in the Treatment of Oral Lichen Planus: A Randomized Controlled Trial.
Brief Title: Evaluation of Efficacy of Neem (Azadirachta Indica) Versus Triamcinolone Acetonide in the Treatment of Oral Lichen Planus.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Goa Dental College (Other Government)
Responsible Party: Principal Investigator, Medhana Mangaonker, Principal Investigator, Goa Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDCH/IEC/I-2024(04)
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-02

CONDITIONS: Oral Lichen Planus
Keywords: Oral Lichen Planus; Neem; Triamcinolone acetonide; corticosteroid; clinical trial
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neem (Experimental)
  Interventions: Drug: Neem gel
- Triamcinolone Acetonide (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Neem gel — 1.5% Neem Gel in orabase formulation, twice daily application for 3 months
  Arms: Neem
Drug: Triamcinolone Acetonide — 0.1% oral paste to be applied twice daily for 3 months
  Arms: Triamcinolone Acetonide

SUMMARY:
The goal of this clinical trial is to learn if Neem works to treat Oral Lichen Planus in adults. It will also learn about the safety of Neem in oral lesions. The main questions it aims to answer are:

To compare the efficacy of 1.5% Neem Gel (Azadirachta Indica) versus 0.1% Triamcinolone Acetonide in treatment of Oral Lichen Planus (OLP) as a topical treatment modality for patients with OLP,

Researchers will compare Neem to a corticosteroid (a standard treatment for Oral Lichen Planus) to see if Neem works to treat Oral Lichen Planus.

Participants:

In experimental group were given Neem Gel in Orabase formulations and control group with topical Triamcinolone acetonide oral paste to be used twice every day for 3 months Visit the clinic once every month for checkups.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical & histopathological diagnosis of OLP.
* Patient above 20 years of age.
* Patient willing to participate in the study with informed consent.
* Patient with recalcitrant OLP.

Exclusion Criteria:

* Patient with known allergic reaction to Triamcinolone Acetonide or Neem.
* Patients with lichenoid lesions.
* Patients with associated cutaneous lesions.
* Pregnant or lactating females.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | From enrollment to the end of 3 months
  Burning sensation will be evaluated with Visual Analogue scale
Thongprasom's Score | From enrollment to the end of the 3 months
  clinical severity of lesion
OLP Disease Severity Score | From enrollment to the end of 3 months
  Site, size and severity of lesion

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | From Enrollment to the end of 3 months
  Anxiety and depression evaluation among patients

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral Medicine and radiology, Goa Dental College and Hospital, Bambolim Goa India, Goa, Bambolim, India

IPD SHARING:
Plan to Share IPD: No